CLINICAL TRIAL: NCT07273981
Title: Phase II Clinical Study of Zanidatamab Combined With Chemotherapy as Neoadjuvant Therapy for Locally Advanced HER2-high Expression (IHC3+/2+FISH+) Gastric/Gastroesophageal Junction Adenocarcinoma
Brief Title: Zanidatamab Combined With Chemotherapy as Neoadjuvant Therapy for HER2-high Expression G/GEJC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJ-G/GEJC-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Gastric/Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Zanidatamab Combined with Chemotherapy (Experimental)
  Interventions: Drug: Zanidatamab Combined with Chemotherapy

INTERVENTIONS:
Drug: Zanidatamab Combined with Chemotherapy — Zanidatamab Combined with Chemotherapy as Neoadjuvant Therapy

SUMMARY:
HER2 overexpression is observed in approximately 20% of gastric cancers and gastroesophageal junction (GEJ) cancers, making it a validated target for anti-tumor therapy . In advanced-stage systemic therapy, trastuzumab combined with chemotherapy has demonstrated clinical benefits for HER2-positive gastric and GEJ cancers . However, the combination of trastuzumab and pertuzumab plus chemotherapy did not significantly improve overall survival (OS) compared to trastuzumab monotherapy in HER2-expressed gastric/GEJ cancers .

In neoadjuvant therapy for early-stage or locally advanced gastric cancer, there is currently no standardized perioperative regimen for HER2-positive gastric or GEJ cancers, and effective treatment remains challenging .

Zanidatamab, a humanized bispecific IgG1-like antibody targeting HER2's ECD4 and ECD2 epitopes, exhibits unique enhanced functionality . Phase II studies (NCT03929666) showed that zanidatamab combined with chemotherapy as first-line therapy for HER2-positive advanced gastroesophageal adenocarcinoma (GEA) demonstrated superior survival benefits and durable responses compared to standard therapy (trastuzumab plus chemotherapy) . A Phase III study (HERIZON-GEA-01, NCT05152147) is now underway to further validate its efficacy when combined with chemotherapy ± tislelizumab versus trastuzumab-based chemotherapy .

For previously untreated stage II/III locally advanced gastroesophageal junction adenocarcinoma (cT1-2N+M0, cT3-4aNanyM0) with confirmed HER2 high expression (HER2 3+/2+ FISH+), neoadjuvant zanidatamab combined with chemotherapy (FLOT/SOX/CAPOX) is being explored to evaluate safety and efficacy, potentially offering a new treatment option for HER2-positive GEJ cancers in perioperative settings .

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Histologically/radiologically confirmed Stage II/III (cT1-2N+M0 or cT3-4aNanyM0) Siewert II/III GEJ/gastric adenocarcinoma.
3. HER2-high (IHC 3+/2+FISH+); HER2 2+ requires FISH (no time restriction).
4. Age 18-75, any gender.
5. ECOG 0-1, surgically eligible.
6. Adequate organ function for abdominal surgery.
7. Life expectancy ≥3 months.

Exclusion Criteria:

Exclusion Criteria

1. Unresectable/metastatic (Stage IV) disease.
2. Prior systemic GC therapy.
3. Other malignancies within 5 years (except those with >90% 5-year survival).
4. Cardiopulmonary dysfunction.
5. Major surgery within 4 weeks pre-study.
6. Severe infection within 4 weeks.
7. Prior chemo/targeted therapy.
8. Hypersensitivity to study drugs/excipients/mAbs.
9. Factors impairing oral intake (e.g., ≥Grade 2 dysphagia/chronic diarrhea).
10. Uncontrolled comorbidities affecting compliance/outcomes.
11. Pregnancy/lactation/planned pregnancy.
12. Immunosuppression (>10mg/day prednisone equivalent within 2 weeks).
13. Active HBV (DNA ≥1×10³ copies/mL or ≥200IU/mL), HCV+, or HIV+.
14. Other antitumor trials within 28 days.
15. Other high-risk conditions (e.g., psychiatric disorders) per investigator.
16. Refusal to sign consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate (MPR) | 24 months
  MPR is defined as 10% or fewer viable cancer cells from the resected tumor following neoadjuvant treatment

SECONDARY OUTCOMES:
Pathological complete response rate(pCR) | 24 months
R0 Resection | 24 months
Recurrence Free Survival (RFS) | 5 years
Treatment-Emergent Adverse Events | 24 months

IPD SHARING:
Plan to Share IPD: No